CLINICAL TRIAL: NCT01477853
Title: A Phase III Randomized Clinical Trial to Study the Efficacy and Safety of the Co-administration of Sitagliptin and Atorvastatin in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: A Study of the Co-administration of Sitagliptin and Atorvastatin in Inadequately Controlled Type 2 Diabetes Mellitus (MK-0431E-211)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early by the Sponsor for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431E-211; 2011-003600-20 (EudraCT Number)
Record Dates: First submitted 2011-11-19; First posted 2011-11-23 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Atorvastatin; Metformin; glimepiride; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin/Sitagliptin + Atorvastatin (Experimental): In Phase A, participants received sitagliptin 100 mg plus matching placebo to atorvastatin daily for 16 weeks. Participants continuing to Phase B received sitagliptin 100 mg plus atorvastatin 80 mg plus matching placebo to glimepiride daily for an additional 38 weeks.
  Interventions: Drug: Sitagliptin; Drug: Atorvastatin; Other: Placebo to atorvastatin; Drug: Metformin (open-label); Drug: Glimepiride (open-label); Drug: Placebo to glimepiride
- Atorvastatin/Atorvastatin + Glimepiride (Active Comparator): In Phase A, participants received atorvastatin 80 mg plus matching placebo to sitagliptin daily for 16 weeks. Participants continuing to Phase B received atorvastatin 80 mg plus matching placebo to sitagliptin plus glimepiride daily for an additional 38 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo to sitagliptin; Drug: Metformin (open-label); Drug: Glimepiride (double-blind)
- Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin (Experimental): In Phase A, participants sitagliptin 100 mg plus atorvastatin 80 mg daily for 16 weeks. Participants continuing to Phase B received sitagliptin 100 mg plus atorvastatin 80 mg plus matching placebo to glimepiride daily for an additional 38 weeks.
  Interventions: Drug: Sitagliptin; Drug: Atorvastatin; Drug: Metformin (open-label); Drug: Glimepiride (open-label); Drug: Placebo to glimepiride

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg tablet orally daily
  Other Names: Januvia
  Arms: Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin; Sitagliptin/Sitagliptin + Atorvastatin
Drug: Atorvastatin — Atorvastatin 80 mg tablet orally daily
  Other Names: Lipitor
Other: Placebo to sitagliptin — Placebo to sitagliptin tablet orally daily
  Arms: Atorvastatin/Atorvastatin + Glimepiride
Other: Placebo to atorvastatin — Placebo to atorvastatin tablet orally daily.
  Arms: Sitagliptin/Sitagliptin + Atorvastatin
Drug: Metformin (open-label) — Participant will remain on prestudy dose of metformin tablets (at least 1500 mg daily) throughout entire study.
  Other Names: Glucophage
Drug: Glimepiride (open-label) — Phase A: Glimepiride 1 or 2 mg tablet once daily with breakfast or the first main meal of the day (titrated up to 6 mg/day) for 16 weeks as rescue therapy for randomized participants not meeting specific glycemic goals.
  Other Names: Amaryl
  Arms: Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin; Sitagliptin/Sitagliptin + Atorvastatin
Drug: Glimepiride (double-blind) — Phase B: glimepiride up to 6 mg daily for participants not rescued with open-label glimepiride during Phase A.
  Arms: Atorvastatin/Atorvastatin + Glimepiride
Drug: Placebo to glimepiride — Phase B: placebo to glimepiride tablet orally daily.
  Arms: Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin; Sitagliptin/Sitagliptin + Atorvastatin

SUMMARY:
This two-phase study was to examine if 16 weeks of treatment with sitagliptin in combination with atorvastatin reduces hemoglobin A1C (A1C) and low density lipoprotein cholesterol (LDL-C) from baseline more than atorvastatin alone and sitagliptin alone, respectively. Following a single-blind placebo run-in period, participants were to be randomized to one of three treatment arms (sitagliptin monotherapy, atorvastatin monotherapy, or sitagliptin plus atorvastatin) for 16 weeks (Phase A). During Phase B of the study (Weeks 16 through 54), participants were to receive either sitagliptin plus atorvastatin or glimepiride plus atorvastatin. The primary hypotheses were that after 16 weeks of treatment, sitagliptin in combination with atorvastatin reduces A1C from baseline more than atorvastatin alone, and that atorvastatin in combination with sitagliptin lowers LDL-C from baseline more than sitagliptin alone.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes mellitus
* is a male, or a female who is highly unlikely to conceive
* is currently on monotherapy with metformin (at least 1500 mg/day) for at least 8 weeks
* is not on statin therapy or other lipid-lowering agents for at least 6 weeks

Exclusion Criteria:

* has a history of type 1 diabetes mellitus, ketoacidosis or possibly has type 1 diabetes
* has ever taken a dipeptidyl peptidase IV inhibitor (such as sitagliptin, vildagliptin, alogliptin, or saxagliptin) or a glucagon-like peptide-1 mimetic (such as exenatide or liraglutide), or has required insulin therapy within 12 weeks prior to signing informed consent
* has been on a peroxisome proliferator-activated receptor gamma agonist within the prior 12 weeks
* has been treated with a statin or other lipid-lowering agents, including over the counter supplements of fish oils within 6 weeks
* intends to consume at least 1.2 liters of grapefruit juice per day during the course of the study
* is on or is likely to require treatment with 14 consecutive days or more, or repeated courses of corticosteroids
* is on a weight loss program and not in the maintenance phase or has started a weight loss medication (such as orlistat or sibutramine) within the prior 8 weeks
* has undergone a surgical procedure within the prior 4 weeks
* has a history of myopathy or rhabdomyolysis with any statin.
* has cardiovascular disease
* has New York Heart Association (NYHA) Class III or IV congestive heart failure, inadequately controlled hypertension, a medical history of active liver disease, chronic progressive neuromuscular disorder, is human immunodeficiency virus (HIV) positive, has a clinically significant hematological disorder, uncontrolled endocrine or metabolic disease known to influence glycemic control or serum lipids/lipoproteins, untreated hyperthyroidism or is currently under treatment for hyperthyroidism
* has a history of malignancy within 5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* is pregnant or breastfeeding, or is intending to become pregnant or donate eggs within the projected duration of the study and post-study follow-up period
* uses recreational or illicit drugs or has had a recent history (within the last year) of drug abuse or increased alcohol consumption

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2011-10-24 (Actual); Primary Completion 2012-12-04 (Actual); Study Completion 2012-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431E-211&kw=0431E-211&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: 10 participants were enrolled in the study more than once (at more than 1 study site). Nine participants were enrolled twice and one participant was randomized at 3 different sites. Therefore, data of 10 actual participants (counted as 21 participants due to multiple screening/randomization) were removed from the efficacy analyses.
Groups:
- Sitagliptin/Sitagliptin + Atorvastatin: In Phase A, participants received sitagliptin 100 mg plus matching placebo to atorvastatin daily for 16 weeks. Participants continuing to Phase B received sitagliptin 100 mg plus matching placebo to glimepiride plus atorvastatin 80 mg daily for an additional 38 weeks.
Period: Phase A
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Started | 55 | 56 | 55
Completed | 12 | 11 | 11
Not Completed | 43 | 45 | 44
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Study terminated by sponsor | 37 | 40 | 39
Period: Phase B
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Started | 12 | 11 | 11
Completed | 0 | 0 | 0
Not Completed | 12 | 11 | 11
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Study terminated by sponsor | 12 | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin | Total
Number analyzed (Participants) | 55 | 56 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (9.7) | 56.3 (8.2) | 53.7 (10.0) | 55.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 24 | 75
  Male | 31 | 29 | 31 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 16
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 16 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 16
Population: Full analysis set (FAS) population included all participants who took at least one dose of study medication and had baseline and at least one post-randomization observation for the analysis endpoint.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 15 | 17 | 14
Percent | -1.17 (0.20) | 0.04 (0.31) | -1.01 (0.22)

2. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 16
Description: Percent change from baseline was calculated as the Week 16 value minus the Week 0 value, divided by the Week 0 value ×100%.
Time Frame: Baseline and Week 16
Population: FAS population included all participants who took at least one dose of study medication and had baseline and at least one post-randomization observation for the analysis endpoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | 4.9 (10.4) | -35.7 (7.1) | -38.7 (6.6)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 16
Description: Change from baseline reflects the Week 16 value minus the Week 0 value.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 15 | 18 | 14
mg/dL | -15.7 (6.4) | 22.7 (10.1) | -26.0 (14.0)

4. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | -1.7 (6.2) | -28.3 (4.8) | -25.7 (6.0)

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | -4.8 (6.5) | -32.9 (5.6) | -29.0 (4.6)

6. Secondary Outcome: Percent Change From Baseline in Non-high Density Lipoprotein Cholesterol (Non-HDL-C) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | -1.0 (8.8) | -34.4 (6.7) | -34.6 (6.7)

7. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | -9.9 (8.6) | -28.7 (6.5) | -10.5 (13.5)

8. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 15 | 18 | 14
Percent change | -15.5 (7.2) | -28.6 (6.6) | -10.4 (13.5)

9. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 16 | 18 | 14
Percent change | -0.3 (3.2) | -5.8 (3.5) | 1.5 (6.0)

10. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the investigational product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the investigational product, is also an adverse event. Data presented exclude data following the initiation of glycemic rescue therapy.
Time Frame: Up to 56 weeks (including 2-week follow-up)
Population: All participants as treated population included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 55 | 56 | 55
Participants | 10 | 13 | 13

11. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 10
Time Frame: Up to 54 weeks
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Number analyzed (Participants) | 55 | 56 | 55
Participants | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to 56 weeks including 2-week follow-up (up to 56 weeks for serious adverse events, up to 54 weeks for non-serious adverse events)
Description: All participants as treated population included all randomized participants who received at least 1 dose of study treatment. Serious adverse events include data after the initiation of rescue therapy and non-serious adverse events exclude data after the initiation of rescue therapy.
Arm/Group | Sitagliptin/Sitagliptin + Atorvastatin | Atorvastatin/Atorvastatin + Glimepiride | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 1/55
Other Adverse Events (participants affected / at risk) | 3/55 | 3/56 | 5/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Sitagliptin + Atorvastatin (N=55) | Atorvastatin/Atorvastatin + Glimepiride (N=56) | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin (N=55)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Sitagliptin + Atorvastatin (N=55) | Atorvastatin/Atorvastatin + Glimepiride (N=56) | Sitagliptin + Atorvastatin/Sitagliptin + Atorvastatin (N=55)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor for business reasons. Due to the small number of participants included in the FAS, the results for Phase A and for the overall study should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.